CLINICAL TRIAL: NCT01213355
Title: A Randomized, Double-Blind, Sponsor Unblinded, Placebo Controlled, 5-Way, Crossover Study To Evaluate The Effects Of Single Oral Administrations of PF-05212377 (SAM-760), A 5-HT6 Antagonist, On Scopolamine Induced Deficits In Psychomotor And Cognitive Function In Healthy Young Adults
Brief Title: Scopolamine Challenge Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: B2081009
Record Dates: First submitted 2010-09-16; First posted 2010-10-04 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Healthy
Keywords: Randomized; double-blind; placebo-controlled; 5-way crossover; single oral administrations of PF 05212377; scopolamine induced deficits in healthy subjects
MeSH Terms: interventions — Scopolamine; SAM-760; Donepezil

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Experimental): placebo, plus scopolamine 0.5 mg
  Interventions: Drug: Placebo; Drug: Scopolamine
- PF-05212377 5 mg, plus scopolamine 0.5 mg; (Experimental)
  Interventions: Drug: PF-05212377; Drug: Scopolamine
- PF-05212377 20 mg, plus scopolamine 0.5 mg; (Experimental)
  Interventions: Drug: PF-05212377; Drug: scopolamine
- PF-05212377 60 mg, plus scopolamine 0.5 mg; (Experimental)
  Interventions: Drug: PF-05212377; Drug: scopolamine
- donepezil 10 mg, plus scopolamine 0.5 mg. (Active Comparator)
  Interventions: Drug: Donepezil; Drug: Scopolamine

INTERVENTIONS:
Drug: Placebo — Capsule, single dose, oral, 1 day
  Arms: Placebo
Drug: Scopolamine — injectable subcutaneous formulation, single dose, 1 day
  Arms: Placebo
Drug: PF-05212377 — 5 mg, PF-05212377, capsule, single dose, 1 day
  Arms: PF-05212377 5 mg, plus scopolamine 0.5 mg;
Drug: Scopolamine — injectable subcutaneous formulation, single dose, 1 day
  Arms: PF-05212377 5 mg, plus scopolamine 0.5 mg;
Drug: PF-05212377 — 20 mg, capsule PF-05212377, single dose, 1 day
  Arms: PF-05212377 20 mg, plus scopolamine 0.5 mg;
Drug: scopolamine — injectable subcutaneous formulation, single dose, 1 day
  Arms: PF-05212377 20 mg, plus scopolamine 0.5 mg;
Drug: PF-05212377 — 60 mg PF-05212377, capsule, single dose, 1 day
  Arms: PF-05212377 60 mg, plus scopolamine 0.5 mg;
Drug: scopolamine — injectable sub cutaneous formulation, single dose, 1 day
  Arms: PF-05212377 60 mg, plus scopolamine 0.5 mg;
Drug: Donepezil — Tablet, 10mg, single dose, 1 day
  Arms: donepezil 10 mg, plus scopolamine 0.5 mg.
Drug: Scopolamine — injectable sub cutaneous formulation, single dose, 1 day
  Arms: donepezil 10 mg, plus scopolamine 0.5 mg.

SUMMARY:
It is hypothesized that PF-05212377 (SAM-760) will reverse scopolamine induced cognitive impairments in healthy adults subjects.

DETAILED DESCRIPTION:
Proof of mechanism

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects of non child bearing potential (WONCBP) between the ages of 18 and 55 years, inclusive.
* Body Mass index (BMI) of between 17.5 to 30.5 kg/m2 inclusive; and a total body weight greater than or equal to 50 kg (110 lbs).

Exclusion Criteria:

* Presence or history of any disorder that may prevent the successful completion of the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2011-04; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Groton Maze Learning Task (Total Errors); included in CogState Battery of Tests. | Day 1 at 0, 5, 6, 7, 8, 10 and 12 hours of each period

SECONDARY OUTCOMES:
Detection Task (Speed; included in CogState Test Battery) | Day 1 at 0, 5, 6, 7, 8, 10 and 12 hours of each period
One Card Learning Task (Accuracy of performance; included in CogState Test Battery) | Day 1 at 0, 5, 6, 7, 8, 10 and 12 hours of each period
Continuous Paired Associate Learning Task (Number of errors; included in CogState Test Battery) | Day 1 at 0, 5, 6, 7, 8, 10 and 12 hours of each period
Bond-Lader Visual Analog Scales (included in CogState Test Battery) | Day 1 at 0, 5, 6, 7, 8, 10 and 12 hours of each period
Identification Task (Speed; included in CogState Test Battery) | Day 1 at 0, 5, 6, 7, 8, 10 and 12 hours of each period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Rennes, France

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B2081009&StudyName=Scopolamine%20Challenge%20Study%20